CLINICAL TRIAL: NCT00289068
Title: Determination of Surgical Efficacy and Most Efficient Surgical Parameters for Use With the 2.2, 2.8, and 3.0mm Phacoemulsification Sleeves Used With the Alcon Infinity 1.1mm ABS Flared Tip
Brief Title: Phacoemulsification Sleeves
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: Phacoemulsification Sleeves
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Cataract
Keywords: cataract surgery; phacoemulsification sleeve
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Phacoemulsification Sleeve 2.2mm: Phacoemulsification Sleeve setting 2.2 mm Procedure/Surgery: Phacoemulsification Sleeves surgery
  Interventions: Procedure: Phacoemulsification Sleeve surgery
- Phacoemulsification Sleeve 2.8mm: Phacoemulsification Sleeve setting 2.8 mm Procedure/Surgery: Phacoemulsification Sleeves surgery
  Interventions: Procedure: Phacoemulsification Sleeves surgery
- Phacoemulsification Sleeve 3.0mm: Phacoemulsification Sleeve setting 3.0 mm Procedure/Surgery: Phacoemulsification Sleeves surgery
  Interventions: Procedure: Phacoemulsification Sleeves

INTERVENTIONS:
Procedure: Phacoemulsification Sleeve surgery — Group 2.2 mm surgery setting
  Other Names: Phacoemulsification Sleeve setting 2.2 mm; Procedure/Surgery: Phacoemulsification Sleeves surgery
  Groups: Phacoemulsification Sleeve 2.2mm
Procedure: Phacoemulsification Sleeves surgery — Group 2.8 mm surgery setting
  Other Names: Phacoemulsification Sleeve setting 2.8mm; Procedure/Surgery: Phacoemulsification Sleeves surgery
  Groups: Phacoemulsification Sleeve 2.8mm
Procedure: Phacoemulsification Sleeves — Group 3.0 mm surgery setting
  Other Names: Phacoemulsification Sleeve setting 3.0 mm; Procedure/Surgery: Phacoemulsification Sleeves surgery
  Groups: Phacoemulsification Sleeve 3.0mm

SUMMARY:
Incision size in cataract surgery is related to induced surgical astigmatism, chamber stability, and surgical efficiency. Sleeves of different diameters change the size of the surgical incision and amount of fluid allowed into the eye during the surgical procedure for a given set of surgical parameters. Optimization of surgical parameters requires review of surgical efficiency including: fluid usage, energy usage, and total surgical time. With optimized surgical parameters recommendations can be made to increase the efficiency and safety of cataract surgery.

DETAILED DESCRIPTION:
No scientific data has been presented comparing the surgical efficiency of the 2.2, 2.8, and 3.0 mm diameter phacoemulsification sleeves for the Alcon Infinity 1.1 mm flare abs tip or the changes in surgical parameters which optimize their performance. Fifty patients per sleeve group will undergo standard cataract extraction with documentation of surgical parameters used for each group. The goal of the study is to determine the most efficient surgical settings for each sleeve diameter and determine statistically the surgical parameters which optimize the use of each phacoemulsification sleeve.

Purpose: The goal of the study is to determine the most efficient surgical settings for each sleeve diameter and determine statistically the surgical parameters which optimize the use of each phacoemulsification sleeve.

Design: The study is designed to allow for scientific evaluation and publication of efficiency parameters using phacoemulsification sleeves of 2.2, 2.8, and 3.0 mm. The proposed study is a prospective nonrandomized clinical investigation of 50 patients per sleeve group.

Methods: Data gathered at the time of surgery will include standard surgical parameters including: Total surgical time, total phacoemulsification/torsional time/power, total volume of infusion fluid, aspiration level, and vacuum level. Post-operative data will include: Post-op day one and week three corneal clarity (clear, would edema, central edema), anterior chamber cell seen in a 2mm 16x magnified slit-lamp biomicroscopic view focused in the aqueous humor (Grade 0 = 0 cells, 1 = up to 10 cells, 2 = 10 to 20 cells, 3 = 20 to 30 cells, 4 = too numerous to count), and uncorrected and/or best corrected visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* requiring cataract surgery

Exclusion Criteria:

* n/a

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dean A. McGee Eye Institute
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2006-01; Primary Completion 2006-04 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Total surgical time, fluid volume, energy used to extract the cataract, post-operative cell and flare and corneal clarity | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David Jackson, MD, Principal Investigator — Dean A. McGee Eye Institute
Locations (1):
- Dean A. McGee Eye Institute, Oklahoma City, Oklahoma, United States